CLINICAL TRIAL: NCT03260842
Title: Bio-Repository of High Risk Cohorts for the Early Detection of Pancreas Cancer
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Walter G. Park, M.D., M.S., Principal Investigator, Stanford University
Other Study IDs: IRB-19286
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cyst; Pancreas Disease
Keywords: early detection; biomarkers; pancreas cancer
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Diseases; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Pancreatic Cyst Fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic Cysts: Patients with pancreatic cyst undergoing endoscopic ultrasound and/or surgery who will have bio-specimens collected
  Interventions: Diagnostic Test: Bio-Specimen Collection
- High Risk Individuals: Patients with established family history and/or genetic mutations for Pancreas cancer who will have bio-specimens collected
  Interventions: Diagnostic Test: Bio-Specimen Collection

INTERVENTIONS:
Diagnostic Test: Bio-Specimen Collection — Collection of bio-specimens and observation over time.

SUMMARY:
Bio-repository to collect bio-specimens from patients with 1) pancreatic cysts and 2) patients at high risk, defined by family history and/or genetic mutations, for pancreatic cancer.

DETAILED DESCRIPTION:
Observational study to collect bio-specimens from 2 separate patient cohorts identified to be at high risk for subsequent development of pancreas cancer.

1. Patients diagnosed with a pancreatic cyst undergoing either endoscopic ultrasound or surgery. Bio-specimens collected include pancreatic cyst fluid and blood. These will be collected using a standard operating protocol.
2. Patients defined as a high risk individual for pancreas cancer by family history and/or known genetic mutations. Bio-specimens collected include blood. This will be collected using a standard operating protocol.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 with pancreas cyst
* Older than 18 at high risk for Pancreas cancer

Exclusion Criteria:

* Unable to provide consent
* Not willing to provide bio-specimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk for developing pancreas cancer defined by the presence of a pancreatic cyst and/or family history or genetic mutation for pancreas cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Pancreas Cancer | 5-10 years
  Development of Pancreas Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Walter Park, MD, Principal Investigator — Faculty
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified clinical and demographic variables may be shared and linked to bio-specimens.